CLINICAL TRIAL: NCT00488124
Title: Evaluation of Growth Response in Short Children Suffering From a Disease With Growth Retardation and Treated With Somatropin: A Prospective, Longitudinal Non-randomised, Open, Phase II Study
Brief Title: Growth Response in Short Children Suffering From a Disease With Growth Retardation and Treated With Somatropin
Acronym: ISS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Professor Dr. med. Doerr, Childrens´ hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRA6280030
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Idiopathic Short Stature
Keywords: short stature
MeSH Terms: conditions — Dwarfism | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin (Genotropin® treatment) — 0,035 mg /kg bodyweight of Somatropin per day given by subcutaneous injections through an injection device (GenotropinPEN)

SUMMARY:
Growth hormone therapy will improve the height of short statured children with pathological conditions that lead to growth retardation. Growth hormone therapy will show an increase in height velocity >1 SD compared to pretreatment height velocity. and the therapy will be safe.

DETAILED DESCRIPTION:
Growth hormone (GH, Somatropin, e.g. Genotropin®) is approved in the treatment of children in specific indications. However, besides the benefit in approved indications, a benefit can also be achieved in other pathological conditions that lead to growth retardation. However, because of their relative low frequency and the long duration of GH studies in children, few data or only case reports on GH treatment are available in these conditions. Nevertheless, published data have suggested a benefit of GH treatment in children suffering from some of those diseases and pediatric endocrinologists sometimes request GH treatment for those children to improve growth rate. This protocol is designed to allow such children with severe growth retardation to be treated with GH and will allow those children to be carefully followed-up and finally evaluated at the end of the GH treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Severe growth retardation (< -2,5 height SDS and annual growth velocity (HV SDS) < 0 SD according to Reinken (1992) and parental adjusted target height < -1 SD according to Tanner (1986)
* Chronological age > 4 and < 10 years, prepubertal children; for girls: Tanner breast stage B = 1, for boys: testis volume ≤ 3 ml
* Any disease which is NOT part of the registered indications for GH treatment in Germany
* Written informed consent from both parents and from the patients if she/he is able to receive and understand the information
* GH treatment requested by an expert in pediatric endocrinology

Exclusion Criteria:

* Participation in any other clinical study
* Unable to follow the and/or comprehend the protocol ( e.g. severe mental retardation)
* Previous history of intolerance or hypersensitivity to the study drug
* History of malignancy
* Chromosomal anomalies with increased risk for malignancy

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2005-11; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To show an improvement of height, change in height (SDS) under GH treatment one year after visit 2 (start of GH therapy). | one and two years of observation

SECONDARY OUTCOMES:
To show an increase in height velocity >1 SD compared to pretreatment height velocity, to confirm good clinical and biological safety of GH treatment in these patients (e.g. adverse events, serum IGF-I, fasting blood glucose and insulin) | one and two years of observation period

CONTACTS AND LOCATIONS:
Overall Officials: Helmuth-Günther Doerr, Prof. Dr., Study Chair — Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (13):
- Germany (13):
  - Kinderklinik, Universitätsklinikum der RWTH Aachen, Pauwelsstraße 30, Aachen
  - Klinik u. Poliklinik für Kinder und Jugendliche, Med. Einrichtungen der Universität Köln, Joseph-Stelzmann-Strasse 9, Cologne
  - Klinik und Poliklinik für Kinder und Jugendliche der Technischen Universität Dresden, Fetscherstr. 74, Dresden
  - Klinik für Kinder und Jugendliche, Schwerpunkt Kinder-Endokrinologie und - Diabetologie, Loschgestr. 15, Erlangen
  - Klinik für Päd. Hämatologie, Onkologie und Endokrinologie, Zentrum für Kinderheilkunde, der Universität Duisburg-Essen, Hufelandstrasse 55, Essen
  - Kinder- und Jugendärztin, Pippinplatz 4, Gauting
  - Endokrinologikum Hamburg, Lornsenstrasse 4 - 6, Hamburg
  - Kinderarztpraxis, Brabeckstrasse 153, Hanover
  - Universitätsklinik für Kinder- und Jugendliche, Abt. Kinderheilkunde, Im Neuenheimer Feld 430, Heidelberg
  - Universitätsklinik für Kinder- und Jugendmedizin, Kirrberger Strasse, Homburg/Saar
  - Zentrum für Frauen und Kindermedizin, Liebigstrasse 20 a, Leipzig
  - Klinik für Allgemeine Pädiatrie und Neonatologie, Otto-von-Guericke-Universität Magdeburg, Leipziger Straße 44, Magdeburg
  - Klinik für Kinderheilkunde und Jugendmedizin, Sektion Pädiatrische Endokrinologie, Hoppe-Seyler-Straße 1, Tübingen